CLINICAL TRIAL: NCT01676129
Title: Comparing the Effect of Typical Electrical Stimulation Therapy With Nocipoint Stimulation Therapy on TMD-Related Myofascial Pain
Brief Title: Nocipoint Therapy Versus Standard Physical Therapy Using Electrical Stimulation in Treating Pain From TMJ Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Pain Cure Center, California (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101R104054-TMJ
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular joint disorders; nocipoint; physical therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nocipoint Therapy (Experimental): Nocipoint therapy (NT) follows rules of TENS stimulation in each session, all within the general FDA guidelines of TENS uses. The key points of Nocipoint Therapy include the following:
  * The stimulation pads are located at the skin surface location of the nociceptors of the muscle/tissue in pain (i.e., "Nocipoint")
  * The intensity is set to induce C-fiber response during the stimulation
  * The duration of stimulation (about 1.5-4 minutes for each tissue stimulation)
  * Stimulations for different tissues (muscles, ligaments) are sequenced such that later stimulations will not cause re-injury of previously treated tissues.
  * Patient are instructed not to use the newly recovered muscle/tissue too much for an estimated "rest period" depending on his/her age.
  Interventions: Procedure: Nocipoint Therapy
- Physical Therapy (Active Comparator): Patients in this group will be treated with comprehensive physical therapy program including typical electrical stimulation using a standard transcutaneous electrical nerve stimulation (TENS) device, manual myofascial release and postural correction exercise.
  The application of TENS will follow general physical therapy guidelines, especially for TMD. Manual myofacial release will be applied on orofacial muscles and neck muscles.
  TENS will serve both as a part of the standard of care and as placebo, as the same TENS device is used in both arms.
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Procedure: Nocipoint Therapy
  Other Names: Charles Koo's Pain Cure Therapy
  Arms: Nocipoint Therapy
Procedure: Physical Therapy
  Arms: Physical Therapy

SUMMARY:
The purpose of this study is to measure the effect of nocipoint therapy on patients with temporomandibular joint disorders (TMD) and compare it with the effect of standard electrical stimulation therapy.

DETAILED DESCRIPTION:
The prevalence of temporomandibular disorders (TMD) is about 20% to 60% of dental patients. Most patients suffer from myofascial pain (MFP) subtype of TMD. Analgesics, local muscle injection or oral appliance are often used to treat TMD-related MFP. Patients are also referred to physical therapists frequently. Many physical therapy (PT) modalities and techniques are applied to these patients, including non-invasive transcutaneous electrical nerve stimulation (TENS) using TENS devices. However, the exact application of TENS devices, including the location of the stimulation, duration and intensity of stimulation, is largely decided by physical therapists. Nocipoint Therapy, a unique combination of precise location, duration and intensity of TENS has been found to substantially relieve general myofascial pain and recover the muscle function with lasting effect.

In preliminary observations of clinical applications, Nocipoint Therapy has been found to rapidly and substantially relieve TMD-related MFP within 2-3 sessions of the treatment.

This clinical study compares the effect of Nocipoint Therapy on TMD with that of standard Physical therapy (PT). TENS will be used in the control group both as a part of the standard of care (i.e., PT) and as placebo.

ELIGIBILITY:
Inclusion Criteria:

* 20-65 years old female or male
* Diagnosed as MFP subtype of TMD according to RDC/TMD
* Pain duration over 3 month
* Tender point in masseter
* Asymmetrical pain intensity
* Subsided symptoms of joint inflammation

Exclusion Criteria:

* Traumatic TMD from external impact force
* History of traumatic cervical injury
* Presence of systemic disease
* Fibromyalgia
* Co-interventions for cervical problems or TMD during study period
* Signs of psychosomatic illness
* Unwilling to be randomized

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for pain | Measurements will be taken before and after each session, and at the follow-up, which is about 4 to 6 weeks after the last session
  VAS is measured before each treatment session and at the follow-up:
  1. VAS - overall
  2. VAS - most painful
  3. VAS - when biting hard food
  4. VAS - at maximal mouth opening range (MMO)
  5. VAS of pressure pain- measured at the three most painful pressure points.
  1,2, and 5 are also measured after each treatment session.

SECONDARY OUTCOMES:
Maximal mouth opening range (MMO) | Measurements will be taken before and after each session, and at the follow-up, which is about 4 to 6 weeks after the last session
Quality of Life (QoL) | Measurements will be taken before the first session and at the follow-up.
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Alex YJ Chen, DDS, PHD, Principal Investigator — National Taiwan University; Charles C Koo, PhD, Principal Investigator — National Taiwan University and Pain Cure Center California; Jau-Yih Tsauo, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- See also: Related Info — http://clinicaltrials.gov/ct2/show/NCT01578148?term=pain+cure+center+california&rank=1